CLINICAL TRIAL: NCT00498225
Title: Randomized Phase III Study of Gemcitabine Versus TS-1 Versus Gemcitabine Plus TS-1 in Unresectable Advanced Pancreatic Cancer (With Local Progression or Metastasis)
Brief Title: Phase III of Gemcitabine Vs TS-1 Vs Gemcitabine Plus TS-1 in Pancreatic Cancer
Acronym: GEST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Collaborators: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01023017
Record Dates: First submitted 2007-07-06; First posted 2007-07-09 (Estimated); Last update posted 2012-11-02 (Estimated); Status verified 2012-11

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; titanium silicide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Gemcitabine plus TS-1
  Interventions: Drug: Gemcitabine plus TS-1
- 2 (Experimental): TS-1
  Interventions: Drug: TS-1
- 3 (Active Comparator): Gemcitabine
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine plus TS-1 — Gemcitabine plus TS-1:Gemcitabine was administered i.v. by 1000 mg/m2 at day 1, 8 followed by 2 week rest as 1 course. TS-1 was co-administered orally at 40 mg/m2 twice daily for 14 days with a rest period of 1 week as one course.
  Arms: 1
Drug: TS-1 — TS-1 was administered orally at 40 mg/m2 twice daily for 28 days with a rest period of 2week as one course.
  Arms: 2
Drug: Gemcitabine — Gemcitabine was administered i.v. by 1000 mg/m2 at day 1, 8, 15 followed by 2 week rest as 1 course.
  Arms: 3

SUMMARY:
In patients with unresectable advanced pancreatic cancer, non-inferiority of TS-1 monotherapy and superiority of GEM + TS-1 combination therapy to gemcitabine (GEM) will be verified using survival time.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic carcinoma histologically determined to be adenocarcinoma or adenosquamous carcinoma.
* Advanced unresectable pancreatic (including pancreatic cancer with local progression and recurrent pancreatic cancer).Presence/absence of measurable lesions is not considered. Patients with measurable lesions must undergo diagnostic imaging tests within 28 days before registration.
* Patients with no previous treatment (radiotherapy,chemotherapy etc) for pancreatic cancer, except resection. Intra-operative radiotherapy during resection of pancreatic cancer will be permitted, although registration must occur at least 4 weeks after the radiotherapy. Patients that have undergone preoperative/postoperative adjuvant chemotherapy may be enrolled if relapse is diagnosed beyond week 24 after the final administration (on day 169 when the day following the final day is set as day 1).
* Age: 20 years to 79 years.
* ECOG Performance Status (PS) of 0 or 1.
* Sufficient function of major organs as defined below. (The following criteria are satisfied in laboratory tests conducted within 14 days before registration. Laboratory tests conducted 2 weeks before registration (on the same weekday) will be included.) White blood cell count≥ 3500/mm3 Neutrophil count≥ 2000/mm3 Hemoglobin≥9.0 g/dL Platelet count≥100000/mm3 Total bilirubin≤ 2.0 mg/dL* *≤ 3.0 mg/dL in patients treated by biliary drainage for obstructive jaundice. AST and ALT≤ 150 U/L Serum creatinine≤1.2 mg/dL Creatinine clearance≥50mL/min.** **Measured values will be used if available. Otherwise, values calculated by the Cockcroft-Gault method will be used.Formula for estimation:body weight (kg) x [140 - age (years) / 72 x serum creatinine (mg/dL)] *Estimated value will be multiplied by 0.85 for females.
* Able to take capsules orally.
* No clinically abnormal ECG findings within 28 days (4 weeks)before registration.
* Voluntarily signed the written consent form.

Exclusion Criteria:

* Pulmonary fibrosis or interstitial pneumonia (to be confirmed by chest X-ray within 28 days before enrollment).
* Watery diarrhoea.
* Active infections (e.g. patients with pyrexia of 38°C or greater), excluding viral hepatitis.
* Serious complications (e.g. heart failure, renal failure,hepatic failure, haemorrhagic peptic ulcer, intestinal paralysis, intestinal obstruction or poorly controlled diabetes).
* Moderate or severe (requiring drainage) ascites or pleural effusion requiring treatment.
* Metastasis in the CNS.
* Active double cancer (synchronous double cancer or asynchronous double cancer with disease-free duration of 3 years or less). Carcinoma in situ and lesions of intramucosal carcinoma will not be included in active double cancer and will be permitted for registration.
* Patients under treatment with flucytosine, phenytoin or warfarin potassium.
* Pregnant females, possibly pregnant females, females wishing to become pregnant and nursing mothers. Males that are currently attempting to produce a pregnancy.
* Severe mental disorder.
* Judged ineligible by physicians for participation in the study from a safety viewpoint.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 834 (Actual)
Dates: Start 2007-07; Primary Completion 2011-07 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Over all survival(OS) | every course for first three courses, then every other course

SECONDARY OUTCOMES:
progression-free survival (PFS), response rate (RECIST, if measurable), incidence rate of adverse events, incidence rate of adverse drug reactions, QOL (EQ-5D) | adverse events will be collected during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Takuji Okusaka, MD, Principal Investigator — National Cancer Center Hospital
Locations (12):
- National Cancer Center Hospital, Tokyo, Japan
- Taiwan (11):
  - Chung-Ho Memorial Hospital, Kaohsiung Medical University, No.100, Tzyou 1st Rd., Kaohsiung
  - Chang Gung Memorial Hospital, Kaohsiung, No.123, Ta-Pei Rd., Niao-Sung Hsiang, Kaohsiung Hsien
  - Changhua Christian Hospital, No.135, Nanxiao St., Changhua
  - National Cheng Kung University Hospital, No.138, Sheng Li Road,Tainan
  - China Medical University Hospital, No.2, Yuh-Der Rd.,Taichung
  - Taipei Veterans General Hospital, No.201, Sec. 2, Shih-Pai Road, Taipei
  - Chi Mei Medical Center Liou Ying Campus, No.201, Taikang Village, Liou Ying Township, Tainan
  - Chang Gung Memorial Hospital, Lonkou, No.5, Fu-Hsing Saint Kuei Shan Hsiang, Taoyuan Hsien
  - National Taiwan University Hospital, No.7, Chung San South Road, Taipei
  - Chi Mei Medical Center, No.901, Chung Hwa Rd., Yong Kang City, Tainan
  - Mackay Memorial Hospital, Taipei, No.92, Sec. 2, Zhongshan N. Rd., Taipei

REFERENCES:
- [Background] Burris HA 3rd, Moore MJ, Andersen J, Green MR, Rothenberg ML, Modiano MR, Cripps MC, Portenoy RK, Storniolo AM, Tarassoff P, Nelson R, Dorr FA, Stephens CD, Von Hoff DD. Improvements in survival and clinical benefit with gemcitabine as first-line therapy for patients with advanced pancreas cancer: a randomized trial. J Clin Oncol. 1997 Jun;15(6):2403-13. doi: 10.1200/JCO.1997.15.6.2403. PMID 9196156
- [Background] Ueno H, Okusaka T, Ikeda M, Takezako Y, Morizane C. An early phase II study of S-1 in patients with metastatic pancreatic cancer. Oncology. 2005;68(2-3):171-8. doi: 10.1159/000086771. Epub 2005 Jul 4. PMID 16006754
- [Background] Ueno H, Okusaka T, Ikeda M, Ishiguro Y, Morizane C, Matsubara J, Furuse J, Ishii H, Nagase M, Nakachi K. A phase I study of combination chemotherapy with gemcitabine and oral S-1 for advanced pancreatic cancer. Oncology. 2005;69(5):421-7. doi: 10.1159/000089997. Epub 2005 Nov 25. PMID 16319514
- [Derived] Okusaka T, Miyakawa H, Fujii H, Nakamori S, Satoh T, Hamamoto Y, Ito T, Maguchi H, Matsumoto S, Ueno H, Ioka T, Boku N, Egawa S, Hatori T, Furuse J, Mizumoto K, Ohkawa S, Yamaguchi T, Yamao K, Funakoshi A, Chen JS, Cheng AL, Sato A, Ohashi Y, Tanaka M; GEST group. Updated results from GEST study: a randomized, three-arm phase III study for advanced pancreatic cancer. J Cancer Res Clin Oncol. 2017 Jun;143(6):1053-1059. doi: 10.1007/s00432-017-2349-y. Epub 2017 Feb 16. PMID 28210843
- [Derived] Ueno H, Ioka T, Ikeda M, Ohkawa S, Yanagimoto H, Boku N, Fukutomi A, Sugimori K, Baba H, Yamao K, Shimamura T, Sho M, Kitano M, Cheng AL, Mizumoto K, Chen JS, Furuse J, Funakoshi A, Hatori T, Yamaguchi T, Egawa S, Sato A, Ohashi Y, Okusaka T, Tanaka M. Randomized phase III study of gemcitabine plus S-1, S-1 alone, or gemcitabine alone in patients with locally advanced and metastatic pancreatic cancer in Japan and Taiwan: GEST study. J Clin Oncol. 2013 May 1;31(13):1640-8. doi: 10.1200/JCO.2012.43.3680. Epub 2013 Apr 1. PMID 23547081